CLINICAL TRIAL: NCT03702387
Title: Evaluation of Second Esmarch Application on Intravenous Regional Anesthesia Effectiveness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Tolga Turker, Assistant Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1705426352
Record Dates: First submitted 2018-04-20; First posted 2018-10-11 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Hand Injuries and Disorders; Anesthesia, Local; Upper Extremity Injury
Keywords: IVRA; Bier Block; Esmarch Bandage
MeSH Terms: conditions — Hand Injuries; Disease; Arm Injuries

STUDY DESIGN:
Intervention Model Description: Male and female patients aged 18-100 who need short upper extremity or hand surgery (cases lasting less than 45 minutes) in the outpatient setting will be considered for the study. Exclusion criteria: patients requesting to withdraw from the study and patients with a history of drug abuse or illicitly used controlled drugs or substances within the last year. The study population will be divided into two groups: one group receiving the standard IVRA procedure and one group receiving the modified IVRA procedure (which simply includes the reapplication of the Esmarch bandage after the local anesthetic is administered intravenously). Due to limited information from other intravenous regional anesthesia studies, at least 40 subjects in each group will be needed (at least 80 patients total). Any patient who would like to participate will be included regardless of comorbidities. Any patient who refuses participation will be excluded, and patients may withdraw from the study at any time.
Who Masked: Participant
Masking Description: Patients will be informed that if they participate in the study, there is a chance they might not receive the modified treatment (and instead receive standard treatment) if they are randomized into the control group. Patients will not be told if they are having the modified IVRA procedure to avoid bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients in this group will have standard intravenous regional anesthesia (IVRA) performed before the start of their surgery.
- Esmarch Reapplication Group (Experimental): Patients in this group will have all the standard intravenous regional anesthesia (IVRA) procedures performed before the start of their surgery with one exception: After standard intravenous regional anesthesia (IVRA) is performed, The elastic Esmarch bandage will be reapplied again on the same arm then will be released. then the surgery will be initiated. the only difference between groups is that the Esmarch reapplied group will be applied the esmach two times. First time, at the standard standard intravenous regional anesthesia (IVRA) before the lidocaine injection and second time, after the injection is completed.
  Interventions: Procedure: standard intravenous regional anesthesia (IVRA) with reapplication of esmach

INTERVENTIONS:
Procedure: standard intravenous regional anesthesia (IVRA) with reapplication of esmach — his intervention simply adds one additional step to the standard IVRA procedure: reapplication of the Esmarch bandage after lidocaine has been injected intravenously. Everything else about this experimental procedure is standard of care.
  Arms: Esmarch Reapplication Group

SUMMARY:
Intravenous regional anesthesia is a commonly used technique in the outpatient setting for short hand and upper extremity cases, such as carpal tunnel release or trigger finger release. The technique requires a tourniquet, Esmarch bandage, an intravenous line, and lidocaine. It can be performed and learned easily. The technique is safe and easy to perform, and it provides adequate anesthesia for short cases; however, there are still some cases in which adequate anesthesia is not achieved. One of the possible reasons for failure is that the local anesthetic (lidocaine) does not properly exit the veins to reach the interstitial space (where many nerves are located) to provide the nerve block. In this study, the investigators hypothesize that after application of lidocaine to the intravenous system, application of external pressure through the skin will facilitate tissue penetration and improve the block. The only research procedure being done is a re-application of the Esmarch bandage; all other procedures are Standard of Care.

DETAILED DESCRIPTION:
Intravenous regional anesthesia (IVRA), also known as Bier block, is a technically simple and reliable technique for achieving anesthesia for short surgical procedures. It is performed by injecting a local anesthetic (usually lidocaine) intravenously in the setting of a double tourniquet on the upper arm which limits the anesthetic effect to that portion of the body to avoid systemic effects. This technique is suitable for short procedures on the forearm and the hand with minimal complications. Variations of the technique alter the location of the tourniquet, the volume of local anesthetic, or the addition of additional anesthetic agents in an effort to provide the best anesthesia. Despite these variations, the block may still fail. Some studies show a success rate of 94-98% while others show a success rate of 78.1% depending on the definition of success (usually defined by whether or not additional anesthesia was necessary during the surgery). In general, however, IVRA has a high success rate. This study aims to improve the success rate (defined by no additional anesthetic needs during surgery) of IVRA by slightly modifying the IVRA protocol. This modification is described in greater detail below (in the research procedures section), but in essence one of the steps involved in the IVRA procedure is to apply an elastic bandage (Esmarch bandage) to the upper extremity to achieve exsanguination before inflating the double tourniquet. The only modification the investigators are making in this study is to reapply the Esmarch bandage in the exact same fashion after the anesthetic has been injected intravenously. This reapplication of the bandage is not for exsanguination but instead for promoting anesthetic extravasation into the interstitial space. Studies show that the main site of action for IVRA is in the interstitial space where small nerve endings and nerve trunks are located. The modification proposed in this study hopes to improve extravasation of the local anesthetic from the venous system into the interstitial space where it will be better able to function. In this study the investigators hope to compare success rates of the standard technique of IVRA to our method in which the investigators reapply the Esmarch bandage soon after injecting local anesthetic intravenously for short hand and upper extremity cases.

Two groups of human subjects with similar demographics will be used for this research: 40 patients randomly assigned to the control group and 40 patients randomly assigned to the study group. The REDCap randomization module will be used for the randomization process, and this process will take place in clinic on the day the patient is recruited and consented. For patients willing to be part of the study, it will be made absolutely clear to them during the consent process that there is a chance they will be assigned to the control group.

In the pre-operative area on the day of the procedure, patients will be reminded of their voluntary participation in the study (and their ability to withdraw at any time before or after the surgery). At this time the individual who initially recruited/consented the patient (e.g. Dr. Turker or Dr. Morin, henceforth "surgeon") will have the patient fill out the demographic information portion of the Bier Block Research Data Collection Form which includes the following: date of birth, sex, BMI, forearm circumference measured at greatest circumference, and comorbidities. Next, the surgeon will fill out the procedure information section of the data collection form which includes the following: date of the procedure, name of the surgeon, name of the anesthesiologist, name of the procedure, and the side of the procedure. At this point the patient may proceed to surgery.

Intravenous anesthesia will be performed using a tourniquet, Esmarch bandage, an intravenous line, and lidocaine diluted with normal saline. First, intravenous access will be obtained on the surgical side, preferably on the dorsum of the hand (however it is standard procedure to try the wrist or forearm if adequate intravenous access cannot be achieved on the dorsum of the hand). Then, a double tourniquet will be applied to the upper arm. An Esmarch bandage will be applied from the fingertips to the tourniquet with protection of the intravenous line. The distal cuff of the tourniquet will then be inflated to 250-300 mmHg. The proximal cuff will be immediately inflated to the same pressure and the Esmarch bandage will be removed. The patient's radial pulse will be checked and the surgeon will then assess the arm for adequate exsanguination prior to injection of 0.5-1% lidocaine, 25-50 milliliters, depending on patient size and anesthesiologist choice. At this point, if the patient was randomized to the study group, the Esmarch bandage will then be applied again in the exact same fashion as above and then immediately removed (this is the ONLY research portion of the study). If the patient was randomized to the control group, the reapplication of the Esmarch bandage will be skipped. Next, the distal cuff will be deflated and the intravenous line on the surgical side will be removed. Standard surgical preparation will commence while the Bier block sets up. If the patient experiences tourniquet pain, the distal cuff will be inflated and the proximal cuff will be deflated. The time to adequate block will be recorded on the data collection form once the patient is no longer able to feel sharp sensation (typically tested by gently poking skin with a sharp surgical instrument). If at any point during the surgery the patient requires additional anesthesia to control pain, the Bier block will be considered a failure. Once adequate pain control is achieved, the surgery proceeds in the usual fashion. Only cases lasting less than 45 minutes will be included in the study. The remainder of the data collection form will be filled out by the surgeon at the end of the procedure and includes the following information: tourniquet time/pressure, block success/failure, blood pressure at time of tourniquet, whether the Esmarch was applied twice, anesthesia type/dose, anatomical IV placement, complications, and additional anesthesia requirements. These completed data collection forms will then be immediately stored in a locked cabinet in the Human Movement Biomechanics Lab (B103). Every week these forms will be transferred to REDCap, and the hard copies will be destroyed securely.

To reiterate and emphasize, the reapplication of the Esmarch bandage is the only research procedure. All other procedures are standard of care. This step may improve the time to adequate block and quality of anesthesia.

After the data from each of the 80 patients' collection forms have been transferred to REDCap, the research team will review and statistically analyze the data. The duration of participation for patients is the length of surgery (in operating room time).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-100.
* Short upper extremity or hand surgery (cases lasting less than 45 minutes).
* Must be outpatient surgery.

Exclusion Criteria:

* Patients requesting to withdraw from the study.
* Patients with a history of drug abuse or illicitly used controlled drugs or substances within the last year.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
IVRA Block Success Rate | This outcome measure will only be measured for the duration of the surgical procedure.
  This study hopes to compare the intravenous regional anesthesia (IVRA) block success rate between the experimental and control groups. The success rate will be defined as whether or not additional anesthesia is needed before or during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Tolga Turker, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Memis D, Turan A, Karamanlioglu B, Pamukcu Z, Kurt I. Adding dexmedetomidine to lidocaine for intravenous regional anesthesia. Anesth Analg. 2004 Mar;98(3):835-40, table of contents. doi: 10.1213/01.ane.0000100680.77978.66. PMID 14980948
- [Background] Brown EM, McGriff JT, Malinowski RW. Intravenous regional anaesthesia (Bier block): review of 20 years' experience. Can J Anaesth. 1989 May;36(3 Pt 1):307-10. doi: 10.1007/BF03010770. PMID 2720868
- [Background] Acalovschi I, Cristea T, Margarit S, Gavrus R. Tramadol added to lidocaine for intravenous regional anesthesia. Anesth Analg. 2001 Jan;92(1):209-14. doi: 10.1097/00000539-200101000-00040. PMID 11133629
- [Background] Dunbar RW, Mazze RI. Intravenous regional anesthesia: experience with 779 cases. Anesth Analg. 1967 Nov-Dec;46(6):806-13. No abstract available. PMID 6070172
- [Background] Lai YY, Chang CL, Yeh FC. The site of action of lidocaine in intravenous regional anesthesia. Ma Zui Xue Za Zhi. 1993 Mar;31(1):31-4. PMID 7968326